CLINICAL TRIAL: NCT04355936
Title: Telmisartan for Treatment of COVID-19 Patients: an Open Label Randomized Trial
Brief Title: Telmisartan for Treatment of COVID-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: Carlos R. Rojo, MD (Unknown); Facultad de Medicina, Universidad de Buenos Aires, UBA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: COVID-19 Drug Treatment
Keywords: COVID-19; TELMISARTAN; ARDS
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive standard care or standard care plus Telmisartan 80 mg twice daily upon diagnosis of COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELMISARTAN (Experimental): Patients in this group will receive 80 mg Telmisartan twice daily plus standard care.
  Interventions: Drug: Telmisartan arm will receive 80 mg Telmisartan twice daily plus standard care.
- CONTROL (No Intervention): Patients in this group will receive standard care.

INTERVENTIONS:
Drug: Telmisartan arm will receive 80 mg Telmisartan twice daily plus standard care. — Control arm will receive standard care.
  Arms: TELMISARTAN

SUMMARY:
In late 2019, a new coronavirus emerged in Wuhan Province, China, causing lung complications similar to those produced by the SARS coronavirus in the 2002-2003 epidemic. This new disease was named COVID-19 and the causative virus SARS-CoV-2. The SARS-CoV-2 virus, enters the airway and binds, by means of the S protein on its surface to the membrane protein ACE2 in type 2 alveolar cells. The S protein-ACE2 complex is internalized by endocytosis leading to a partial decrease or total loss of the enzymatic function ACE2 in the alveolar cells and in turn increasing the tissue concentration of pro-inflammatory angiotensin II by decreasing its degradation and reducing the concentration of its physiological antagonist angiotensin 1-7. High levels of angiotensin II on the lung interstitium can promote apoptosis initiating an inflammatory process with release of proinflammatory cytokines, establishing a self-powered cascade, leading eventually to ARDS. It has recently been proposed the tentative use of agents such as losartan and telmisartan as alternative options for treating COVID-19 patients prior to development of ARDS. The present study is an open-label randomized phase II clinical trial for the evaluation of telmisartan in COVID-19 patients. Briefly, patients with confirmed diagnosis of SARS-CoV-2, will be randomized to receive 80 mg/12h of telmisartan plus standard care or standard care alone aand will be monitored for development of systemic inflammation and acute respiratory distress syndrome. Other variables regarding lung function and cardiovascular function will also be evaluated.

DETAILED DESCRIPTION:
In late 2019, a new coronavirus emerged in Wuhan Province, China, causing lung complications similar to those produced by the SARS coronavirus (SARS-CoV) in the 2002-2003 epidemic. This new disease was named COVID-19 and the causative virus SARS-CoV-2 (Chen, Liu, & Guo, 2020; Li et al., 2020).

Given that vaccines against COVID-19 are still in development and an effective treatment against this new coronavirus is lacking, various pharmacological agents are being tested in clinical trials designed by institutions such as the WHO or scientific entities in different countries (C.-C. Lu, Chen, & Chang, 2020).

Taking into account the characteristics of the mode of entry of this coronavirus to human cells through binding with Angiotensin Converting Enzime 2 (ACE2) and extensive scientific and clinical evidence information on the Renin Angiotensin System, the hypothesis of the involvement of this system in the pathophysiology of COVID-19 was born (Gurwitz, 2020; Vaduganathan et al., 2020).

The SARS-CoV-2 virus, enters the airway and binds, by means of the S (Spike) protein on its surface (after whose image the term coronavirus is coined), to the membrane protein ACE2 in type 2 alveolar cells (R. Lu et al., 2020; Wan, Shang, Graham, Baric, & Li, 2020). The S protein-ACE2 complex is internalized by endocytosis and facilitates the entry of each virion into the cytoplasm. For each intracellular entry, the function of one ACE2 molecule is lost leading to a partial decrease or total loss of the enzymatic function ACE2 in the alveolar cells of the lung directly related to the viral load of the air inoculum.

ACE2 catalyzes the transformation of angiotensin II into angiotensin 1-7. Angiotensin II acting on AT1 receptors causes vasoconstriction, apoptosis, proinflammatory effects, and fibrosis. Angiotensin 1-7 acting on Mas receptors causes opposite effects: vasodilation and anti-inflammatory. Partial decrease or total loss of ACE2 function in alveolar cells results in a deviation of the homeostatic balance of the Renin Angiotensin System in favor of the angiotensin II-AT1 receptor axis (Paz Ocaranza et al., 2020; Tikellis, Bernardi, & Burns, 2011). Indeed, it increases the tissue concentration of angiotensin II by decreasing its degradation and reduces the concentration of its physiological antagonist angiotensin 1-7(Liu et al., 2020).

The clinical manifestations of COVID-19 disease will depend fundamentally on the degree of alteration of the homeostatic balance of the Renin Angiotensin System in the lung and at the systemic level (mainly at the heart).

Increasing the effects of angiotensin II on the lung interstitium can promote apoptosis, which, in turn, initiates an inflammatory process with release of proinflammatory cytokines, establishing a self-powered cascade (Cardoso et al., 2018). In certain patients this process reaches such clinical relevance that requires external oxygen supply and in severe cases an Acute Respiratory Distress Syndrome (ARDS) ensues (this correlates with an acute release -storm- of cytokines) (Ware & Matthay, 2000).

Based on the aetiopathogenic hypothesis described, there are various pharmacotherapeutic proposals to be evaluated through clinical trials: Recombinant ACE2 therapy, administration of agents aimed at increasing ACE2 levels (e.g. estradiol), and administration of drugs that decrease the elevated activity of angiotensin II including renin release inhibitors, classic ACE inhibitors or Angiotensin Receptor 1 Blockers (ARBs).

Most patients who develop COVID-19 disease initially have fever, indicative ofan inflammatory process with systemic release of pyrogenic cytokines. According to the hypothesis described, this inflammation is induced by the inhibition of ACE2 and the imbalance of the renin angiotensin system in the pulmonary interstitium in favor of the angiotensin II-AT1 receptor axis. Faced with the onset of the inflammatory process, a rapidly effective treatment is necessary to antagonize the cascading and self-sustaining phenomenon described. Of the different types of drugs mentioned above, we consider that the most rapidly effective may be ARBs.

Recently, Gurwitz (2020) proposed the tentative use of agents such as losartan and telmisartan as alternative options for treating COVID-19 patients prior to development of ARDS.

ARBs are widely used to treat hypertension and there is an abundant clinical experience with its use, all representatives of this group being characterized by their excellent tolerance; Furthermore, its adverse effects profile has been described as "placebo like(Schumacher & Mancia, 2008; Sharpe, Jarvis, & Goa, 2001).

The most suitable ARB to antagonize the proinflammatory effects of angiotensin II in a patient with a recent positive COVID-19 test should be the compound with the best pharmacological properties for this indication. From the comparative analysis of the available ARBs, telmisartan gathers properties that make it the best pharmacological tool to evaluate the hypothesis under discussion in a clinical trial.

Liposolubility is relevant for absorption after oral administration and for tissue penetration. Telmisartan stands out among all the representatives of the ARBs for being markedly more lipophilic, expressed both in partition coefficients (octanol / neutral pH buffer), distribution coefficients and distribution volumes (Vd). Telmisartan has a Vd of approximately 500 L, irbesartan 93 L, and both valsartan and olmesartan, candesartan and losartan, approximately 17 L.

The affinity of ARBs for the AT1 receptor has been measured by multiple studies, mainly using radioligand binding studies. All AT1 receptor blockers are characterized by having similar affinity values (pKi or pIC50, between 2 and 19 nM), with losartan and its active metabolite EXP3174 being the lowest and irbesartan, candesartan and telmisartan the highest (Kakuta, Sudoh, Sasamata, & Yamagishi, 2005).

Using isolated organ technique on blood vessels from different tissues and from different animals, these AT1 antagonists have a blocking power (pA2) against angiotensin II in the nM range (losartan, 8.15; irbesartan, 8.52; valsartan, 9.26; telmisartan 9.48; candesartan, 10.08). Telmisartan has a 10-fold higher blocking potency than losartan (Kakuta et al., 2005).

Functional as well as biochemical studies determining the dissociation rates of the ARBs have shown that these drugs have a slow dissociation rate that gives them characteristics of pseudo-irreversible blocking agents. In the only comparative study using cloned human AT1 receptors, the half-lives of receptor dissociation were: telmisartan, 213 min; olmesartan, 166 min; candesartan, 133 min; valsartan, 70 min; losartan, 67 min (Kakuta et al., 2005). Telmisartan is the AT1 blocker that dissociates more slowly from the receptor. This property may be clinically relevant as it maintains a longer lasting blockade difficult to reverse by the endogenous agonist angiotensin II.

Furthermore, telmisartan causes downregulation of AT1 receptor at the mRNA and protein level apparently due to its action as a partial agonist of PPAR-gamma (Peroxisome Proliferator-Activated Receptor gamma). This action can contribute to the effects of telmisartan by producing a decrease in the number of AT1 receptors (Imayama et al., 2006).

In summary, telmisartan, which is well absorbed after oral administration, is the ARB with the longest plasma half-life (24 h), it reaches the highest tissue concentrations due to its high lipid solubility and high volume of distribution (500 L), and dissociates more slowly after binding to the AT1 receptor, causing an apparently irreversible block (Kakuta et al., 2005; Michel, Foster, Brunner, & Liu, 2013).

The present study is an open-label randomized phase II clinical trial for the evaluation of telmisartan in COVID-19 patients. Briefly, patients with confirmed diagnosis of SARS-CoV-2, will be randomized to receive 80 mg/12h of telmisartan (Bertel®, Laboratorio Elea Phoenix, Buenos Aires, Argentina) plus standard care or standard care alone will be monitored for development of systemic inflammation and acute respiratory distress syndrome. Other variables regarding lung function and cardiovascular function will also be evaluated.

Clinical studies to evaluate the safety of Telmisartan in healthy individuals or in hypertensive patients with daily doses of up to 160 mg, found no difference between those treated with telmisartan and the placebo group in frequency and intensity of adverse effects (Schumacher & Mancia, 2008; Sharpe et al., 2001; Stangier, Su, & Roth, 2000).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed diagnosis of COVID-19 by PCR test
* Hospitalization for COVID-19
* Illness symptoms beginning 4 days or less prior to randomization

Exclusion Criteria:

* Admitted to ICU prior to randomization
* Illness symptoms beginning more than 4 days prior to randomization
* Pregnancy
* Breast feeding
* Major hypersensibility to angiotensin receptor blockers (ARBs)
* Systolic blood pressure < 100mmHg
* Potassium greater than 5.5 mEq/L
* AST and/or ALT > 3 times the upper limit of normal
* Serum creatinine higher than 3 mg/dL
* Current treatment with angiotensin converting enzyme inhibitor (ACEi) or ARB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
C reactive protein | Days 5 and 8 after enrollment
  Serum C rective protein levels

SECONDARY OUTCOMES:
Admission to intensive care unit (ICU) | Within 15 and 30 days after randomization
Occurrence of mechanical ventilation | Within 15 and 30 days after randomization
Death | Within 15 days and 30 days
  All-cause mortality; and time to all-cause mortality
Composite occurrence of admission to ICU, mechanical ventilation or death (what occur first) | Within 15 and 30 days after randomization
Time from randomization to discharge | Within 15 days
Proportion of patients not requiring supplemental oxygen at day 15 | Within 15 days
Significative differences in serum lactate dehydrogenase | Days 5 and 8
  Troponin serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Azzato, MD, Study Chair — Department of Internal Medicine, Hospital de Clínicas 'José de San Martín', Facultad de Medicina, Universidad de Buenos Aires; Mariano Duarte, MD, Principal Investigator — Hospital de Clínicas 'José de San Martín', Universidad de Buenos Aires
Locations (2):
- Argentina (2):
  - Hospital de Clínicas 'José de San Martín', Facultad de Medicina, Universidad de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Hospital Español de Buenos Aires, Buenos Aires

REFERENCES:
- [Derived] Duarte M, Pelorosso F, Nicolosi LN, Salgado MV, Vetulli H, Aquieri A, Azzato F, Castro M, Coyle J, Davolos I, Criado IF, Gregori R, Mastrodonato P, Rubio MC, Sarquis S, Wahlmann F, Rothlin RP. Telmisartan for treatment of Covid-19 patients: An open multicenter randomized clinical trial. EClinicalMedicine. 2021 Jun 18;37:100962. doi: 10.1016/j.eclinm.2021.100962. eCollection 2021 Jul. PMID 34189447
- [Derived] Rothlin RP, Vetulli HM, Duarte M, Pelorosso FG. Telmisartan as tentative angiotensin receptor blocker therapeutic for COVID-19. Drug Dev Res. 2020 Nov;81(7):768-770. doi: 10.1002/ddr.21679. Epub 2020 May 1. PMID 32356926